CLINICAL TRIAL: NCT02097511
Title: A Randomized, Open-label, Three-sequence, Three-period Crossover Study to Investigate The Effect of Anplag on the Disposition of Betaloc in Healthy Male Volunteers
Brief Title: Sarpogrelate Drug Interaction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Doo-Yeoun Cho, Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DDI-102
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Hypertension; Peripheral Artery Disease
Keywords: Drug-drug interaction; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Hypertension; Peripheral Arterial Disease | interventions — sarpogrelate; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sarpogrelate pretreatment and Metoprolol (Experimental): Sarpogrelate hydrochloride 100 mg pretreatment three times a day for three days and Metoprolol Tartrate 100 mg once a day with Sarpogrelate hydrochloride 100 mg three times a day
  Interventions: Drug: Sarpogrelate pretreatment; Drug: Sarpogrelate; Drug: Metoprolol
- Sarpogrelate and Metoprolol (Active Comparator): Metoprolol Tartrate 100 mg once a day with Sarpogrelate hydrochloride 100 mg three times a day
  Interventions: Drug: Sarpogrelate; Drug: Metoprolol
- Metoprolol only (Active Comparator): Metoprolol Tartrate 100 mg once a day
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Sarpogrelate pretreatment — Sarpogrelate hydrochloride 100 mg pretreatment three times a day for three days
  Arms: Sarpogrelate pretreatment and Metoprolol
Drug: Sarpogrelate — Sarpogrelate hydrochloride 100 mg three times a day
  Arms: Sarpogrelate and Metoprolol; Sarpogrelate pretreatment and Metoprolol
Drug: Metoprolol — Metoprolol Tartrate 100 mg once a day

SUMMARY:
This is a randomized, open-label, single & multiple-dose, three-sequence, three-period crossover study to investigate the effect of sarpogrelate hydrochloride on the disposition of metoprolol tartrate in healthy male volunteers

DETAILED DESCRIPTION:
Eligibility for participation of this study will be determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 4 weeks before study drug administration. Subjects suitable for this study will be admitted to the Clinical Trial Center of Ajou University Medical Center on the day before dosing (Day -1).

On Day 1, Subjects will be dosed study drug (metoprolol tartrate 100 mg once a day only, or metoprolol tartrate 100 mg once a day with sarpogrelate hydrochloride 100 mg three times a day, sarpogrelate hydrochloride 100 mg three times a day pretreatment for three days and metoprolol tartrate 100 mg once a day with sarpogrelate hydrochloride 100 mg three times a day).

Pharmacokinetic samplings and blood pressure/pulse rate measurement will be done upto 12 hours after metoprolol tartrate 100 mg dosing.

After one week of washout period (Day 8), Subjects will be dosed study drug by crossover manner, and pharmacokinetic samplings and blood pressure/pulse rate measurement will be done upto 12 hours after metoprolol tartrate 100 mg dosing.

After one week of washout period (Day 15), Subjects will be dosed study drug by crossover manner, and pharmacokinetic samplings and blood pressure/pulse rate measurement will be done upto 12 hours after metoprolol tartrate 100 mg dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 45 years
* With in 20% of ideal body weight, {Ideal body weight=[height(cm)-100]*0.9}
* Agreement with written informed consent

Exclusion Criteria:

* Clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal disease or mental disorder (Past history or present)
* Inadequate result of laboratory test (especially, AST/ALT > 1.25 x UNL, Total bilirubin > 1.5 x UNL)
* Positive reaction in the HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL test
* Taking OTC(Over the counter)medicine including oriental medicine within 7 days
* Clinically significant allergic disease (Except for mild allergic rhinitis and dermatitis seems to be not need for medication)
* Subject with known for hypersensitivity reaction to Metoprolol or Sarpogrelate
* Previous whole blood donation within 60 days or component blood donation within 30 days
* Previous participation of other trial within 90 days
* Continued taking caffeine (caffeine > 5 cup/day), drinking (alcohol > 30 g/day) and severe heavy smoker (cigarette > 1/2 pack per day)
* An impossible one who participates in clinical trial by investigator's decision including for reason of laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Metoprolol and metabolites | upto 12 hours after Metoprolol Tartrate 100 mg dosing
  Cmax (maximal plasma concentration) and AUC (area under the time-concentration curve) will be calculated from pharmacokinetic samplings

SECONDARY OUTCOMES:
Blood pressure and pulse rate changes | Upto 12 hours after Metoprolol Tartrate 100 mg dosing
  Blood pressure and pulse rate measurement with Dash 5000 patient monitoring system (GE Healthcare, USA) at 0 (before Metoprolol Tartrate 100 mg dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12 hours after Metoprolol Tartrate 100 mg dosing

CONTACTS AND LOCATIONS:
Overall Officials: Doo-Yeoun Cho, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea